CLINICAL TRIAL: NCT03418948
Title: Comparison of Adenoma Miss Rate and Adenoma Detection Rate Between Endocuff Vision®-Assisted Colonoscopy and Conventional Colonoscopy: a Multicenter Randomized Trial
Brief Title: Comparison of AMR and ADR Between Endocuff Vision-assisted and Conventional Colonoscopy: a Multicenter Randomized Trial
Acronym: EXCEED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Norgine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: EXCEED study
Record Dates: First submitted 2017-12-18; First posted 2018-02-01 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2017-12

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants will be blinded for the allocation. Physicians can not be blinded for the use of Endocuff, but during the first procedure they will be blinded for the second procedure method to limit observer related bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 2 x CC (Active Comparator): 2 x conventional colonoscopy (CC), back-to-back design
  Interventions: Device: 2x CC
- CC followed by EC (Active Comparator): Conventional colonoscopy followed by Endocuff Vision- assisted colonoscopy, back-to-back design
  Interventions: Device: CC followed by EC
- EC followed by CC (Active Comparator): Endocuff Vision-assisted colonoscopy followed by conventional colonoscopy, back-to-back design
  Interventions: Device: EC followed by CC
- 2 x EC (Active Comparator): 2 x Endocuff Vision-assisted colonoscopy
  Interventions: Device: 2x EC

INTERVENTIONS:
Device: CC followed by EC — CC = conventional colonoscopy EC = endocuff assisted colonoscopy
  Arms: CC followed by EC
Device: EC followed by CC — CC = conventional colonoscopy EC = endocuff assisted colonoscopy
  Arms: EC followed by CC
Device: 2x EC — EC = endocuff assisted colonoscopy
  Arms: 2 x EC
Device: 2x CC — CC = conventional colonoscopy
  Arms: 2 x CC

SUMMARY:
The aim of this international multicenter study is to compare the adenoma detection rate and adenoma miss rate of conventional and Endocuff Vision-assisted colonoscopy.

DETAILED DESCRIPTION:
Rationale: Population screening programs for colorectal cancers (CRC) are increasingly adapted as a public health initiative with the primary goal to prevent CRC and CRC related deaths. [2-4] The ultimate benefit of CRC screening relies on the detection and resection of (pre-)malignant colon lesions, and for this colonoscopy is the preferred modality. Recently, concerns have been raised about the effectiveness of colonoscopy in the prevention of CRC after several studies reported unexpected high incidence rates of interval carcinomas (IC), especially in the proximal colon.[5-9] Most ICs are suspected to arise from missed colon lesions during colonoscopy. The retrograde approach of colonic inspections may contribute to colon lesions remaining undetected as it limits visualization of the proximal sides of haustral folds and flexures. Endocuff Vision® is a single-use, disposable medical device designed to improve the detection of colon lesions. The 'finger-like' projections of the device provide fold retraction allowing the visualization of otherwise hidden anatomical areas. Additionally, Endocuff Vision® may improve scope tip stability and prevent scope slippage.

Objectives:

1. To compare adenoma miss rates (AMR) between Endocuff Vision®-assisted colonoscopy (EAC) and conventional colonoscopy (CC)
2. To compare adenoma detection rates (ADR) between EAC and CC
3. To assess whether a proposed increased ADR and reduced AMR with EAC is indeed due to the fold-flattening device or merely a consequence of the second colonoscopy procedure performed.
4. To assess the clinical relevance of the polyps missed during the first colonoscopy procedure.

Study design: This multicenter, randomized, same-day, back-to-back tandem colonoscopy trial will include four separate study groups: group A; CC followed by CC, Group B; CC followed by EAC, Group C; EAC followed by CC, and group D; EAC followed by EAC.

Study population: Patients between the ages of 40 and 75-years referred for screening (non-IFOBT based), diagnostic or surveillance colonoscopy.

Main study parameters/endpoints: The primary endpoint of the study will be AMR.

Secondary endpoints include; ADR, mean number of adenomas detected per colonoscopy procedure, number of sessile serrated polyps, the total number of colon lesions found during the first and second examination (which will be compared for size, colon distribution, morphologic and histopathological characteristics), cecal intubation rates, bowel cleansing levels, procedure times, sedation use, (severe) adverse events, patient reported outcome (pain) and post-colonoscopy surveillance intervals applying European and United states surveillance guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Patients, aged between 40 and 75-years old, referred and scheduled for either screening (non-FIT/gFOBT based), diagnostic or surveillance colonoscopy.

Exclusion Criteria:

* Prior surgical resection of any portion of the colon or a history of radiotherapy for any abdominal or pelvic disease.
* Personal history of colon cancer or polyposis syndrome.
* Familial adenomatous polyposis (FAP)
* Known colitis or suspicion of colitis (ulcerative colitis, Crohn's colitis, diverticulitis, infective colitis).
* Lower gastro-intestinal bleeding requiring acute intervention.
* Suspicion of large bowel obstruction or toxic megacolon.
* Prior incomplete colonoscopy (not including insufficient preparation).
* Patients referred for a therapeutic procedure or assessment of a known non-resected lesion.
* Not sufficiently corrected anticoagulation disorders
* Poor general condition (>3 American Society of Anesthesiologist)
* Overweight (>120 kg)
* Inability to provide informed consent.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 708 (Estimated)
Dates: Start 2017-12-08 (Actual); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
Adenoma miss rate (%) | 18 months
  To compare adenoma miss rates (AMR) between Endocuff Vision®-assisted colonoscopy (EAC) and conventional colonoscopy (CC)

SECONDARY OUTCOMES:
Adenoma detection rate (%) | 18 months
  To compare adenoma detection rates (ADR) between Endocuff Vision®-assisted and CC.
Mean number of adenomas detected per colonoscopy procedure | 18 months
  Mean number of adenomas detected per colonoscopy procedure. This will be calculated after the first and second procedure to assess if there is a significant increase.
Number of sessile serrated lesions per procedure | 18 months
  Number of sessile serrated lesions per procedure. This will be calculated after the first and second procedure to assess if there is a significant increase.
Total number of colon lesions found during first and second examination | 18 months
  These polyps will be compared for size, colon distribution (coecum, ascending, transversum, descending, sigmoïd or rectum), morphologic (Paris classification) and histopathological characteristics (Vienna classification)
Difference in ADR (learning curve first 20% and last 20% by each colonoscopist) | 18 months
  To compare the ADR of the first 20% of patients scoped by each colonoscopist with the last 20% of patients in each arm to identify any changes in ADR throughout the trial (to assess a learning curve) between CC and EC
Cecal intubation rate | 18 months
  To compare cecal intubation rates between both techniques.
Bowel cleansing levels; using the Boston Bowel Preparation Scale (BBPS) ranging from 0-9) | 18 months
  To compare BBPS scores between both techniques. A BBPS score of 2 or more in each colon segment is considered adequate.
Procedure times (minutes) | 18 months
  To compare procedure times; total procedure time, insertion time, mean polypectomy time, withdrawal time)
Number of severe adverse events | 18 months
  To compare the number of severe adverse events between study groups. 1 month follow-up
Sedation and analgesia use; type and amount | 18 months
  To compare the use of sedation and analgesia between study groups. Type of sedation and analgesia and amount will be compared
Post-polypectomy surveillance guidelines; difference in surveillance intervals after the first and second procedure. | 18 months
  To compare post-colonoscopy surveillance intervals applying European and US surveillance guidelines.
To compare patient reported outcomes e.g. pain | 18 months
  Visual Analog Scale 2 days and 1 month after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Peter D Siersema, MD, Principal Investigator — Radboud University Medical Center
Locations (3):
- Greece (2):
  - "Attikon" University General Hospital,, Athens, Haidari
  - 417 Army Veterans Hospital, Athens
- Radboud University Medical Center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van Keulen KE, Papanikolaou IS, Mak TWC, Apostolopoulos P, Neumann H, Delconte G, Furnari M, Peters Y, Lau JYW, Polymeros D, Schrauwen RWN, Cavalcoli F, Koukoulioti E, Triantafyllou K, Anderson JC, Pohl H, Rex DK, Siersema PD. Comparison of adenoma miss rate and adenoma detection rate between conventional colonoscopy and colonoscopy with second-generation distal attachment cuff: a multicenter, randomized, back-to-back trial. Gastrointest Endosc. 2024 May;99(5):798-808.e3. doi: 10.1016/j.gie.2023.11.017. Epub 2023 Nov 20. PMID 37993062